# Study protocol

Assessment of intercostal block scheduling in preventing acute surgical and post-surgical pain in thoracoscopic surgery

Entrepreneur : Dr. Dan Levy Faber

Address: Medical cente Carmel St. Michel 7, Haifa, 34362

Site of the study: Department Surgery chest House Patients Carmel

Principle Investigator: Dr. Dan Levy Faber

# **Protocol Summary:**

Background: Patients undergoing Thoracic surgery may suffer from postoperative severe pain. Today there is widespread use of the minimally invasive approach called VATS = video assisted thoracoscopic surgery. This approach reduces postoperative pain, but pain balance is still a Controversial issue. In most surgeries performed in our unit, an intercostal block, with Bupivacaine, is given during surgery to relieve postoperative pain. This study examines whether the timing of block performance at the beginning or end of the surgery affects the quality of the patient's pain control balance.

Methods: This study is a prospective comparative clinical trial between two groups of patients. Each group will include 30 randomly assigned patients with similar demographic characteristics. Patients were recruited from the surgical community in the Department of Chest Surgery at Carmel Medical Center according to the inclusion criteria.

In the study group, an intercostal block will be performed at the beginning of the operation and in the control group the intercostal block will be performed at the end of the operation.

The follow-up of Patients will include: assessment of pain levels in the days after surgery using visual analogue scale (VAS), calculation of the amount of pain medication intake during hospitalization, duration of hospitalization, and surgical and postoperative complications.

Study participants will be above 18 years old and able to sign an informed consent.

## Inclusion Criteria

Above 18 years old

Thoracoscopic Surgery

No Known allergy to kamacaine

Able to sign an informed consent

#### Non inclusion Criteria

Previous surgery in the same side of the thorax

## Inter costal BUPIVACAINE block

Is an analgesic procedure the involve the injection of BUPIVACAINE between the ribs close the intercostal nerve. This procedure blocks the pain transmission of the nerves

BUPIVACAINE Is an anesthesia medicine from the Amino-amides Family. It is being used for many years the action of the drug Based On tying of The material To the sodium canals voltage dependent within the cells and blocking the passage of the sodium to the nerves cells. This block prevents depolarization of The cells. No cell Depolarization meaning No pain.

The purpose of the experiment:

The study try to appreciate the quality of pain control during and after thoracoscopic surgery and to see whether change in the timing of the intercostal block improve pain control

## REFERENCE

.1 Regional analgesia for video-assisted thoracic surgery: a systematic review.Steinthorsdottir KJ, Wildgaard L, Hansen HJ, Petersen RH, Wildgaard K. Eur J Cardiothorac Surg. 2013 Nov 27.

.2 Postoperative analgesia in video-assisted thoracoscopy : the role of intercostal blockade. Taylor R, Massey S, Stuart-Smith K .

| J Cardiothorac Vasc Anesth . 2004 Jun ; 18 (3): 317-21 . |
|---|
| . 3 The efficacy of intraoperative inner intercostal nerve block during video-assisted thoracic surgery on postoperative pain.Bolotin G, Lazarovici H, Uretzky G, Zlotnick AY, Tamir A, Saute M.Ann Thor ac Surg. 2000 Dec; 70 (6): 1872-5. |
| . 4 Preventing post-thoracotomy pain syndrome.Khelemsky Y, Noto CJ . |
| Mt Sinai J Med. 2012 Jan-Feb ; 79 (1): 133-9. doi : 10.1002 / msj.21286.<br>Review . |
| .5 Prevention of chronic pain after surgical nerve injury: amputation and thoracotomy.Buchheit T, Pyati S.Surg Clin North Am. 2012 Apr ; 92 (2): 393-407. Review . |
| . 6 Paravertebral blocks.Chelly JE. Anesthesiol Clin . 2012 Mar ; 30 (1): 75-90. Review . |

. 7 Persistent postoperative pain: where are we now? Niraj G, Rowbotham  $\operatorname{DJ}$  .

Br J Anaesth